CLINICAL TRIAL: NCT06598449
Title: Assessment of Safety of the Use of Fenfluramine in Children With Dravet Syndrome Under the Age of 24 Months
Brief Title: Assessment of Safety of the Use of Fenfluramine in Children With Dravet Syndrome Under 24 Months of Age
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-3972
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Dravet Syndrome (DS); Children Under 2 Years
Keywords: Fenfluramine; Dravet Syndrome; Children under 2 years
MeSH Terms: conditions — Epilepsies, Myoclonic | interventions — Fenfluramine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fenfluramine (Experimental): The dose of FENFLURAMINE for the duration of the Treatment Period will range from 0.2 mg/kg/day to a maximum of 0.7 mg/kg/day, not to exceed a total daily dose of 26 mg/day; for patients concurrently being prescribed stiripentol, the maximum will be 0.4 mg/kg/day, not to exceed a total daily dose of 17 mg/day.
  Under this treatment plan, FENFLURAMINE will be administered twice daily in equally divided doses, with at least 8 hours and no more than 12 hours between doses in a single day.
  Interventions: Drug: fenfluramine

INTERVENTIONS:
Drug: fenfluramine — Clear, cherry flavored oral solution

SUMMARY:
Dravet syndrome is a genetic epilepsy associated with pathogenic variants in SCN1A that codes for Nav1.1, a protein necessary for sodium channels. Children with Dravet syndrome classically present in the first year of life with prolonged seizures, often hemiclonic and in the setting of fever or temperature changes such as getting in or out of bath water. Many anti-seizure medications are sodium channel blockers and exacerbate seizures in this patient population. This creates some limitations in medication choices for this patient population. Recently fenfluramine was approved for use in Dravet syndrome for people 2 years and older. Randomized studies demonstrated a 74.9% reduction of convulsive motor seizures compared to 19.2% in the placebo group. Additionally, 16% of children treated with fenfluramine were seizure free. Fenfluramine is likely to be as effective in children under the age of 2 years. The current study has proposed a treatment protocol to allow access to fenfluramine for children under 24 months of age.

ELIGIBILITY:
Inclusion Criteria:

Treating physicians must submit a clinical statement of potential benefit to the lead site for review of the multi-PIs, which includes patient's gender, age, diagnosis, genetic pathogenic variant, co-morbidities, seizure history, prior and current therapies, response to prior therapies and reason for request. Echocardiogram (ECHO) results must also be submitted to the lead site prior to final approval. Patients must be between 12 and 23 months old to be eligible. Each subject will be reviewed by the multi-PIs to ensure agreement that the subject has Dravet syndrome. Additional inclusion criteria:

1. SCN1A with a known or presumed pathogenic variant or VUS with a history of prolonged seizure or a clinical diagnosis of Dravet syndrome.
2. Failure of at least one anti-seizure medication that is not a sodium channel blocker (lamotrigine, oxcarbazepine, carbamazepine, eslicarbazepine)

Exclusion Criteria:

1. Patients with mild or greater mitral valve regurgitation and/or trace or greater aortic valve regurgitation will not be eligible for participation. The clinical statement can be submitted first for initial, conditional approval and then ECHO results can be submitted at a later date for final approval.
2. Patients with failure to thrive will not be eligible for participation as fenfluramine can suppress appetite and has a risk for weight loss. Failure to thrive will be evaluated on the following criteria:

   1. Weight less than the 2nd percentile.
   2. Lack of weight gain that crosses two or more of the major percentile lines and is not congruent with length.

Inclusion of patients will be at the sole discretion of the multi-PIs based on a majority vote.

Ages: 12 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants that have at least one adverse event | 12 months
  A description of the percentage of participants that have at least one adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Knupp, MD, Principal Investigator — University of Colorado, Denver; Joseph Sullivan, MD, Principal Investigator — University of California, San Francisco; Elaine Wirrel, MD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - University of California San Francisco, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: Undecided